CLINICAL TRIAL: NCT01758263
Title: Economic Impact of Switching From Metoprolol to Nebivolol for Hypertension Treatment: A Retrospective Database Analysis
Brief Title: Economic Impact of Switching From Metoprolol to Nebivolol for Hypertension Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: NEB-HE-200
Record Dates: First submitted 2012-12-26; First posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-12

CONDITIONS: Hypertension
Keywords: Hypertension; Health Care Cost; Monthly health care cost
MeSH Terms: conditions — Hypertension | interventions — Metoprolol; Nebivolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metoprolol to Nebivolol: Patients with high blood pressure (hypertension) who were continuously treated with metoprolol for a minimum of 6 months prior to switching to nebivolol. Patients were then continuously treated with nebivolol for a minimum of 6 months.
  Interventions: Drug: Metoprolol; Drug: Nebivolol

INTERVENTIONS:
Drug: Metoprolol — Metoprolol, oral administration
Drug: Nebivolol — Nebivolol, oral administration

SUMMARY:
This is a retrospective data analysis of patients with high blood pressure (hypertension) who took metoprolol for a minimum of 6 months who then switched to taking nebivolol for a minimum of 6 month to treat hypertension. These patients will be identified from a large medical claims database. This study tests the hypothesis (alternative, higher or lower) that average patient monthly health care administrative cost changes after switching from metoprolol to nebivolol.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old at initiation of metoprolol (or first date on metoprolol treatment between 2007 and 2011)
* Had one or more inpatient or outpatient claims with a primary or non-primary diagnosis of hypertension (ICD-9-CM 401.xx-405.xx)
* Received nebivolol treatment continuously (defined as supply gap <30 days) for at least 6 months after initiation
* Received metoprolol treatment continuously for at least 6 months prior to switching to (initiation of) nebivolol (defined as metoprolol was discontinued whereas a prescription for nebivolol was filled)
* Had at least 12 months of continuous enrollment (as verified using enrollment file): 6 month prior to nebivolol initiation and 6 months following nebivolol initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patents treated for hypertension during the period of 2007-2011 in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2012-10; Primary Completion 2012-12 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Patient monthly health care cost | 6 months
  The average per patient monthly health care cost for the pre-specified hypertensive target study population during the 6 months before and after switching from metoprolol to nebivolol

SECONDARY OUTCOMES:
Number of monthly out-patient visits | 6 months
  Estimate the average per patient monthly number of out-patient visits for the pre-specified hypertensive target study population during the 6 months before and after switching from metoprolol to nebivolol.
Monthly Emergency Room visits per patient | 6 months
  Estimate of the average monthly number of Emergency Room (ER) visits per patient for the pre-specified hypertensive target study population during the 6 months before and after switching from metoprolol to nebivolol.
Monthly hospitalizations per patient | 6 months
  Estimate of the average monthly number of hospitalizations per patient for the pre-specified hypertensive target study population during the 6 months before and after switching from metoprolol to nebivolol.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Chen, PhD, Study Director — Forest Laboratories
Locations (1):
- Forest Investigative Site 0, Jersey City, New Jersey, United States